CLINICAL TRIAL: NCT03294668
Title: Developing and Evaluating a Social Skills Group Training for Adolescents on the Autism Spectrum
Brief Title: KONTAKT Australia a Social Skills Group Training for Adolescents on the Autism Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Curtin University (Other)
Collaborators: Autism Association of Western Australia (Unknown); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Sonya Girdler, Associate Professor, Curtin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRE2017-0245
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Autism Spectrum Disorder
Keywords: social skills group training; Adolescents; Active control group; Australian
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The participants will be randomly allocated into an intervention group (KONTAKT Australia) and an active control group (Social cooking group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The Assessor is blind to the participant's allocation to the intervention and active control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KONTAKT Australia (Experimental): A social skills group training
  Interventions: Behavioral: KONTAKT Australia
- Super Chef (Active Comparator): A social cooking group
  Interventions: Other: Super Chef

INTERVENTIONS:
Behavioral: KONTAKT Australia — KONTAKT is a manualized Social skills group training program designed for children and adolescents on the Autism Spectrum aimed at improving communication, social interaction skills, the severity of ASD symptoms, and the ability to empathise and adapt in a group setting. The KONTAKT participants (4-8 participants) meet face to face weekly for 16 weeks for an hour and a half in a group facilitated by two trainers.
  Other Names: KONTAKT
  Arms: KONTAKT Australia
Other: Super Chef — The Super Chef is a cooking group designed for this study for adolescents on the Autism Spectrum, aimed at teaching basic cooking skills in a social environment. The Super Chef participants (4-8 participants) meet face to face weekly for 16 weeks for an hour and a half in a group facilitated by two trainers.
  Other Names: Social cooking group
  Arms: Super Chef

SUMMARY:
This study evaluates the KONTAKT social skills group training in Australian adolescents on the autism spectrum compared to an active control group which is a group cooking class

DETAILED DESCRIPTION:
KONTAKT is a manualized Social Skills Group Training program designed for children and adolescents with ASD which aims to improve communication, social interaction skills, reduce the severity of ASD symptoms, improve the ability to empathise and adapt in a group setting. A large randomized controlled trial in Sweden found that adolescents who participated in KONTAKT demonstrated improvements in social skills, behaviour, reduced stress and improved overall functioning as reported by parents immediately following and at three months after the program. However, social skills are at least in part influenced by social cultural contexts and there is a need to understand the feasibility, acceptability and effectiveness of KONTAKT in an Australian context. Moreover, in the previous studies, the social skills groups were compared to treatment as usual groups. Therefore, this study evaluates the KONTAKT social skills group training in Australian adolescents on the autism spectrum compared to an active control group which is a group cooking class

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 12 to 17
* Clinical consensus diagnosis of ASD as defined by DSM-5 and confirmed by the Autism Diagnostic Observation schedule-2
* IQ scores > 70 as measured by the Wechsler Abbreviated Scale of Intelligence - Second Edition (WASI-II)

Exclusion Criteria:

* Existing prior comorbid externalizing behaviours as assessed by the Childhood Behaviour Checklist (CBCL).
* Clinically assessed self-injurious behaviour
* Low intrinsic motivation to participate in a social skills training group
* Insufficient English language skills

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-10-06 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Change in the Goal Attainment Scale (GAS) | Baseline (week 0), Post-test (week 20), follow up (week 36), and long follow up (week 74)
  The GOAL Attainment Scale will be used as the adolescents' primary outcome. Using the scale the participants personally meaningful social goals will be specified, and a behavioural expectation that ranges from the worst to the best possible outcome will be listed for each goal. This allows qualitative data to be quantified in relation to the success of the participant in achieving expectations of change.

SECONDARY OUTCOMES:
Change in the Emotion Regulation and Social Skills Questionnaire (ERSSQ) | Baseline (week 0), Post-test (week 20), follow up (week 36), and long follow up (week 74)
  The parents will fill this questionnaire (Parent form). This is a 27-item measure assessing emotion regulation and competency in social skills.The questionnaire is designed to measure frequencies of effective engagement in social behaviours (e.g. "chooses appropriate solutions to social problems" or "deals effectively with bullying"), examining the competency of these skills. Responses are rated on a 5-point Likert scale, ranging from "never (0)" to "always (4)", yielding a total score of 0-108, with higher scores indicating higher competencies in social behaviour.
Mind Reading Battery | Baseline (week 0), Post-test (week 20) and follow up (week 36)
  The adolescents will fill this questionnaire. Emotions are displayed in the form of 2-5 second silent coloured video clips, with 4 multiple choice options one of which is the correct emotion label and 3 are distractor items. The distracter options were randomly selected from the entire Mind reading battery emotion groups, excluding the emotion group the target stimuli originates from. Further details of the stimuli are outlined in table 4. During the presentation of stimuli, eye tracking data will be recorded via a Remote Eye Tracker Device (RED) developed by SensoMotoric Instruments, enabling examination of fixation patterns and fixation durations.
Change in the Circumplex Scale of Interpersonal Efficacy (CSIE) | Baseline (week 0), Post-test (week 20) and follow up (week 36)
  The adolescents will fill this questionnaire. It measures an individual's confidence in regard to their ability to successfully perform behaviours associated with each facet of the interpersonal Circumplex (Assert, Distance, Yield, and Connect). Each octant scale shows a progressive blend of two axial dimensions (e.g. "speak up" representing an assertive action, "get them to leave me alone" a distancing action, and "tell them when I am annoyed" combining these two actions).
Change in the Paediatric Quality of life Inventory- 4th edition (PedQL-4.0) | Baseline (week 0), Post-test (week 20) and follow up (week 36)
  The adolescents and parents (parent proxy) both will fill this questionnaire. It is a 23-item parent proxy report and an adolescent self-report measure of adolescent's quality of life underpinned by the four subscales of physical, emotional, social, and school functioning. Responders rate items according to if they have been a problem for them on a 5-point Likert scale ranging from "never (0)" to "almost always (5)", with lower scores indicating better quality of life.
Change in the Perth Loneliness Scale (PALs) | Baseline (week 0), Post-test (week 20), follow up (week 36), and long follow up (week 74)
  The adolescents will fill this questionnaire. This is a self-report measure consisting of 24 statements such as ''I feel left out of things at school'', or ''I get along with my classmates'', measuring four dimensions of loneliness in young people (isolation, friendship and positive and negative attitudes toward solitude).
Change in the Negative Incidents and Effects of Psychological Treatment (NEQ) | Post-test (week 20) and follow up (week 36)
  The adolescents will fill this questionnaire. The NEQ is a 32-item questionnaire requiring adolescents to quantify, on 5-point Likert scale with response options ranging from "Not at all" to "Extremely", any negative events experienced during the intervention period, asking participants to attribute their causality to either the program or external circumstances
Change in the Child Health Utility 9D (CHU9D) | Baseline (week 0), Post-test (week 20), follow up (week 36), and long follow up (week 74)
  The adolescents will fill this questionnaire. This is a 9-dimension Health related quality of life scale (worried, sad, pain, tired, annoyed, school work, sleep, daily routines and activities), designed to estimate the adolescent's Quality adjusted life years (QALY), providing a standardized measure of disease burden. The measure is rated on a 5-point scale with a "don't" sentence linked with no problems (e.g. I don't feel sad today) and "very" with the participant experiencing a lot of problems (e.g. I feel very sad). Calculation of an universal score is supported by an adolescent specific scoring algorithm, with 1 representing 'full health' and 0 'death'.
Change in Emotions via Experience Sampling (ESM) | Through the intervention until follow up time from week 1 to 36
  The adolescents and parents (parent proxy) will fill this questionnaire. This 5-item measure, specifically designed for the purposes of this study, asks "In the last 24 hours, on a scale of 1 to 10 I have been feeling …" with answers rated on a 10-point scale regarding five dichotomised emotional sets (sad/happy, lonely/unlonely, angry/calm, scared/unafraid, and anxious/confident).
Change in Social Interaction Anxiety Scale (SIAS) | Baseline (week 0), Post-test (week 20), follow up (week 36), and long follow up (week 74)
  The adolescents will fill this questionnaire. This is a 20-item measure assessing adolescents' self-reported anxiety in social situations, via items such as "I become tense if I have to talk about myself" or "I find it easy to make friends my own age". Items are rated on a 5-point scale ranging from "Not at all" to "extremely". Total scores range from 0 to 80 with higher scores indicating greater anxiety in social situations
Change in Treatment Inventory of Costs in Patients (TIC-P) | Baseline (week 0), Post-test (week 20), follow up (week 36), and long follow up (week 74)
  The parents will fill this questionnaire (Parent form). This will be measured via a tailored version of the Trimbos/iMTA questionnaire for patients with a psychiatric disorder (TiC-P), a well-established questionnaire examining health care usage as well as any work, education and productivity losses incurred by participants and their carers. The modified version of the TIC-P employed in this study comprise six sections enquiring about health care visits, support received both at and outside of school, medications and supplements, work, and education and productivity losses incurred by both parents and adolescents.
Change in social functioning | Time 1 (week 3), Time 2 (week 13 ), Time 3 (week 19)
  This will be assessed by a blinded assessor
Treatment Satisfaction Scale | Post-test (week 20)
  The adolescents and parents both will fill this questionnaire. This is a short 6-item parent and adolescents self-report instrument, measuring satisfaction with group attendance. Each item is scored on a 4-point Likert scale with response options ranging from "Yes, very much" to "No" with an open comment section, encouraging participants to freely share their experiences with the intervention.
Change in the Social responsiveness scale - Second Edition (SRS-2) | Baseline (week 0), Post-test (week 20), follow up (week 36), and long follow up (week 74)
  This measure will be used as the parent's primary outcome.The Social Responsiveness Scale - Second Edition (SRS-2) School-Age Form is a 65-item rating scale, designed to measure social deficits in individuals with ASD via parent proxy report has been used as the primary outcome in a previous study evaluating KONTAKT and has been used as the basis for the power calculation for the present RCT.

CONTACTS AND LOCATIONS:
Overall Officials: Sonya J Girdler, PhD, Principal Investigator — Occupational Therapy Professor - Curtin University
Locations (1):
- Curtin University, Bentley, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afsharnejad B, Falkmer M, Black MH, Alach T, Lenhard F, Fridell A, Coco C, Milne K, Chen NTM, Bolte S, Girdler S. Cross-Cultural Adaptation to Australia of the KONTAKT(c) Social Skills Group Training Program for Youth with Autism Spectrum Disorder: A Feasibility Study. J Autism Dev Disord. 2020 Dec;50(12):4297-4316. doi: 10.1007/s10803-020-04477-5. PMID 32270385
- [Background] Afsharnejad B, Falkmer M, Black MH, Alach T, Lenhard F, Fridell A, Coco C, Milne K, Chen NTM, Bolte S, Girdler S. KONTAKT(c) for Australian adolescents on the autism spectrum: protocol of a randomized control trial. Trials. 2019 Dec 9;20(1):687. doi: 10.1186/s13063-019-3721-9. PMID 31815642
- [Background] Afsharnejad B, Falkmer M, Picen T, Black MH, Alach T, Fridell A, Coco C, Milne K, Perry J, Bolte S, Girdler S. "I Met Someone Like Me!": Autistic Adolescents and Their Parents' Experience of the KONTAKT(R) Social Skills Group Training. J Autism Dev Disord. 2022 Apr;52(4):1458-1477. doi: 10.1007/s10803-021-05045-1. Epub 2021 May 3. PMID 33942186
- [Result] Afsharnejad B, Falkmer M, Black MH, Alach T, Lenhard F, Fridell A, Coco C, Milne K, Bolte S, Girdler S. KONTAKT(R) social skills group training for Australian adolescents with autism spectrum disorder: a randomized controlled trial. Eur Child Adolesc Psychiatry. 2022 Nov;31(11):1695-1713. doi: 10.1007/s00787-021-01814-6. Epub 2021 May 30. PMID 34052908